CLINICAL TRIAL: NCT02810145
Title: The Incidence and Magnitude of Cerebral Desaturation in Traumatic Brain Injury (TBI) Patients
Brief Title: Cerebral Desaturation in Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Duane Funk, Associate Professor, University of Manitoba
Other Study IDs: HS19659
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Brain Injuries
Keywords: traumatic brain injury; cerebral desaturation; intensive care; hemodynamics; Loss; Consciousness
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TBI with GCS <or= 8: Adult patients admitted to the surgical intensive care unit with traumatic brain injury and a Glasgow coma score less than or equal to 8.

SUMMARY:
We will determine the incidence and magnitude of cerebral desaturation in TBI. Adult patients (18 years and older) admitted to the Surgical/Trauma Intensive Care Unit (ICU) at the Health Sciences Center with a severe TBI will have cerebral oximetry monitoring instituted within 12 hours of admission and continuing for 72 hours after placement. Decreases in regional cerebral oxygenation will be correlated with ICU hemodynamic parameters including mean arterial pressure, intracranial pressure, and arterial oxygen and carbon dioxide tension.

DETAILED DESCRIPTION:
In patients who have suffered a traumatic brain injury, the current management strategies focus on the maintenance of normotension and normoxia and a normalized intracranial pressure (ICP). Recent evidence calls into question the utility of ICP monitoring in these patients. More advanced cerebral monitoring such as the use of invasive brain tissue oxygen monitors have not found their way into widespread clinical practice. Cerebral oximetry monitoring utilizes the different absorption characteristics of oxygenated and deoxygenated blood to measure global brain oxygen levels.

While clinicians have no ability to reverse the primary brain injury, they can mitigate the secondary injury effects, namely hypoxia and hypotension. It is well known that maintaining normal blood pressure and oxygen saturation can prevent secondary brain injury. However, it is also known that despite the appearance of normal hemodynamics, brain oxygen delivery in the ischemic penumbra may be inadequate. This secondary brain injury is likely related to decreases in cerebral oxygenation (rSO2).

There have been a number of studies that have examined a link between intraoperative decreases in rSO2 and adverse perioperative outcome. These studies suggest that decreases in rSO2 may be related to both adverse neurologic and non-neurologic sequelae. All of these studies suffer from similar flaws, however. They are typically small in size, have varying definitions of what constitutes a cerebral desaturation event, and have incompletely, or poorly defined complications. Also lacking is a mechanistic explanation for the cerebral desaturations as peripheral oxygen saturation typically remains near normal.

The brain can be considered the organ of highest priority when it comes to tissue hypoperfusion during shock states. When oxygen delivery to the brain is decreased below a critical value, cerebral desaturations occur. In the context of TBI, cerebral desaturation may be the hallmark of secondary injury. Consistent with this hypothesis, in the largest cerebral oximetry trial to date, Murkin and colleagues discovered that the incidence and magnitude of cerebral desaturations was related to major non-neurologic organ morbidity.

Two questions arise in relation to this prior research. First, are these cerebral desaturations causative of the adverse outcomes, and second if these desaturations were treated (i.e. if cerebral oxygenation was normalized) would outcome be improved (i.e. or are cerebral desaturations merely an epiphenomenon)?

This study will determine the incidence and severity of cerebral desaturation in traumatic brain injury patients admitted to the Surgical Intensive Care Unit. We will examine factors associated with cerebral desaturation such as ICP and blood pressure, and will determine if decreases in rSO2 are helpful in prognostication of traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older admitted to ICU with severe TBI (Glasgow coma score <or=8)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Surgical/Trauma ICU at Health Sciences Centre, Winnipeg with a severe TBI (Glasgow coma score < or = 8).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of cerebral desaturation | 72 hours
  The frequency of cerebral desaturation from time of admission to 72 hours post admission to ICU as measured by rSO2 output from cerebral oximetry.
Magnitude of cerebral desaturation | 72 hours
  The magnitude of cerebral desaturation from time of admission to 72 hours post admission to ICU as measured by rSO2 output from cerebral oximetry.

SECONDARY OUTCOMES:
Association between cerebral desaturation and intracranial pressure | 72 hours
  Cerebral desaturation measured by rSO2 output from cerebral oximetry vs intracranial pressure over 72 hours post admission to ICU by an adjusted regression model
Association between cerebral desaturation and mean arterial pressure | 72 hours
  Cerebral desaturation measured by rSO2 output from cerebral oximetry vs mean arterial pressure over 72 hours post admission to ICU by an adjusted regression model
Association between cerebral desaturation and arterial oxygenation | 72 hours
  Cerebral desaturation measured by rSO2 output from cerebral oximetry vs arterial oxygen tension over 72 hours post admission to ICU by an adjusted regression model
Association between cerebral desaturation and arterial carbon dioxide concentration | 72 hours
  Cerebral desaturation measured by rSO2 output from cerebral oximetry vs arterial CO2 over 72 hours post admission to ICU by an adjusted regression model

CONTACTS AND LOCATIONS:
Overall Officials: Duane J. Funk, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer GW. Recent advances in application of cerebral oximetry in adult cardiovascular surgery. Semin Cardiothorac Vasc Anesth. 2008 Mar;12(1):60-9. doi: 10.1177/1089253208316443. Epub 2008 Apr 7. PMID 18397905
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Fischer GW, Lin HM, Krol M, Galati MF, Di Luozzo G, Griepp RB, Reich DL. Noninvasive cerebral oxygenation may predict outcome in patients undergoing aortic arch surgery. J Thorac Cardiovasc Surg. 2011 Mar;141(3):815-21. doi: 10.1016/j.jtcvs.2010.05.017. Epub 2010 Jun 25. PMID 20579669
- [Background] Kazan R, Bracco D, Hemmerling TM. Reduced cerebral oxygen saturation measured by absolute cerebral oximetry during thoracic surgery correlates with postoperative complications. Br J Anaesth. 2009 Dec;103(6):811-6. doi: 10.1093/bja/aep309. PMID 19918024